CLINICAL TRIAL: NCT02715479
Title: A Two-way Drug Interaction Study to Evaluate the Effect of BMS-955176 on the Pharmacokinetics of Dolutegravir and the Effect of Dolutegravir on the Pharmacokinetics of BMS-955176
Brief Title: A Study to Evaluate the Effect of BMS-955176 on Pharmacokinetics of Dolutegravir and the Effect of Dolutegravir on the Pharmacokinetics of BMS-955176
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 206222; AI468-052 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; BMS-955176

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Single DTG tablet under fed conditions for a specified period
  Interventions: Drug: Dolutegravir
- Treatment B (Experimental): Two BMS955176 tablets under fed conditions for a specified period
  Interventions: Drug: BMS955176
- Treatment C (Experimental): Single DTG tablet and Two BMS955176 tablets under fed conditions for a specified period
  Interventions: Drug: Dolutegravir; Drug: BMS955176

INTERVENTIONS:
Drug: Dolutegravir — Dolutegravir
  Arms: Treatment A; Treatment C
Drug: BMS955176 — BMS955176
  Arms: Treatment B; Treatment C

SUMMARY:
The purpose of this study is to evaluate how BMS955176 affects pharmacokinetics (PK) of Dolutegravir (DTG) and also how DTG administration affects the PK of BMS955176

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Target population: Healthy males and females.
3. Women of child bearing potential (WOCBP) with negative serum pregnancy test
4. Women must not be breastfeeding
5. Men and WOCBP must agree to follow instructions for contraception

Exclusion Criteria:

1. History of any chronic or acute illness, gastrointestinal disease, GI surgery, cardiac disease or clinically significant cardiac arrhythmia
2. History of frequent headaches or acute diarrhoea.
3. Any major surgery within 4 weeks of study drug administration
4. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population
5. History of allergy to HIV maturation and integrase inhibitors,or related compounds
6. History of smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) for DTG | Days 1 to 5 and days 15 to 21
Area under the concentration-time curve in 1 dosing interval AUC (tau) for DTG | Days 1 to 5 and days 15 to 21
Maximum observed plasma concentration (Cmax) for BMS-955176 | Days 8-21
Area under the concentration-time curve in 1 dosing interval AUC (tau) for BMS-955176 | Days 8-21

SECONDARY OUTCOMES:
Adverse events (AEs) | Days 1-21; for SAEs up to 30 days post discontinuation of dosing
  The incidence of observed AEs will be tabulated and reviewed for potential significance and clinical importance.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

REFERENCES:
- See also: Description BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: Description Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx
- See also: Description FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/